CLINICAL TRIAL: NCT00837759
Title: Novel Therapy Combining Regenerative Stimuli Immunomodulation to Preserve Beta Cell Function in New Onset Type 1 Diabetes
Brief Title: Novel Therapy to Preserve Beta Cell Function in New Onset Type 1 Diabetes
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Changes to study personnel.
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, James Balow, Clinical Director Intramural NIDDK, National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090056; 09-DK-0056 (Other: National Institutes of Health Clinical Center); 09-DK-0056 (Other: NIHCC)
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Results first posted 2012-10-24 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-12

CONDITIONS: Diabetes Mellitus Type 1; Autoimmune Diabetes
Keywords: Type I Diabetes; Preserve Beta Cell Function; Sitagliptin; Lansoprazole; GAD65 (Diamyd); Diabetes; Type 1 Diabetes; T1DM
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Insulin; Lansoprazole; Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- T1D group (Other): This study was terminated prior to full subject accrual because of changes to study personnel. The original study design was changed from a double-blind, placebo-controlled study to an open-label pilot study in order to collect safety data on enrolled subjects prior to study termination.
  Interventions: Drug: Insulin; Drug: Lansoprazole; Drug: Sitagliptin; Biological: Diamyd; Drug: GAD65 (Diamyd)

INTERVENTIONS:
Drug: Insulin
Drug: Lansoprazole
Drug: Sitagliptin
Biological: Diamyd
Drug: GAD65 (Diamyd)

SUMMARY:
Background:

* Type 1 diabetes (T1D) occurs when the immune system attacks insulin-producing cells (beta cells) in the pancreas, resulting in their death.
* Insulin injections currently are the best method for controlling blood sugar in individuals with T1D. However, animal studies have shown that the drugs sitagliptin and lansoprazole can help reverse beta cell damage or develop new beta cells. In addition, Diamyd has been shown to weaken the immune process that attacks pancreatic beta cells.

Objectives:

* To find out whether a combination treatment of sitagliptin, lansoprazole, and Diamyd will help maintain functioning beta cells and/or cause new beta cells to form.
* To determine how the drug combination affects insulin doses and blood sugar control.
* To determine whether the drug combination affects the immune response involved in T1D.

DETAILED DESCRIPTION:
Type 1 diabetes (T1D) is the end result of immune mediated beta-cell destruction. It is generally accepted that at the time of T1D is diagnosed, an individual has lost most (60-80%) of his/her beta cell function. The loss of insulin-producing beta cells is believed to occur over a period of months to years and individuals can retain some endogenous insulin production even years after clinical diagnosis of diabetes. The presence of residual beta cell mass may signify a complex interplay between the auto-destructive immune response and the capacity for limited beta cell regeneration. When initiated at T1D onset, immunosuppression has been shown to preserve beta cell function, but with significant and limiting toxicities. Selectively targeting the pathogenic T-cells involved in T1D development and progression could achieve the same objective with less toxicity. Various studies of the non-obese diabetic (NOD) mouse model of spontaneous autoimmune diabetes have demonstrated that administering glutamic acid decarboxylase (GAD65), a beta cell autoantigen, can prevent the immune destruction and delay or prevent diabetes onset. Preclinical studies have also identified several growth factors, including epidermal growth factor (EGF), glucagon-like peptide 1 (GLP-1), and gastrin, that appear to promote beta cell proliferation. We seek to test the potential for preserving beta cell function early in the disease course of T1D by combining antigen-specific immunomodulation with regenerative stimuli.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Recently diagnosed (within the preceding 4 months of screening) diabetes clinically consistent with T1D:

     A. Positive for anti-GAD antibody.

     B. BMI between 19 and 28 kg/m2; for those between the ages of 16 to 18, the BMI must be within 10th to 90th percentile for the age.
  2. Ages between 16 and 30 years, inclusive
  3. Random plasma C-peptide level of equal to or greater than 0.20 nmol/L
  4. Willingness and ability to institute intensive insulin-based glucose management.

EXCLUSION CRITERIA:

1. Diabetic nephropathy with a creatinine clearance less than 60 cc/min or 24 hour urine albumin greater than 300 mg
2. Insulin requirements greater than 0.8 units/kg/day at the end of the run-in period
3. Regular use of a proton pump inhibitor within 3 months of enrollment
4. Use of GLP-1R agonist or DPP-4 inhibitor within 6 months prior to enrollment
5. Use of immunosuppressive therapy in the preceding 12 months
6. Evidence of chronic infection, for example, known human immunodeficiency virus (HIV) or hepatitis
7. History of any malignancy other than a treated basal or squamous skin cancer
8. Any chronic medical condition to unduly increase risk for the potential enrollee as judged by study investigators
9. Pregnancy, breastfeeding or planned pregnancy within two years, women of reproductive age not using an effective mode of contraception and unwilling to continue adequate contraception until 1 year after the last study drug administration
10. Any other co-existing condition/circumstances that would make patient unsuitable to participate in the study, as deemed by the investigators. For example, study investigators would exclude any potential candidate with any of the following (but the list is not inclusive):

A. Clinically significant past history of an acute reaction to vaccines or other drugs

B. Recent participation in other clinical trials with a new chemical entity

C. A history of alcohol or drug abuse

D. Significant neurological conditions like epilepsy, head trauma, or cerebrovascular accidents

E. Individuals with significant gastrointestinal disorders determined by the study investigators to influence either study safety or data interpretation. Such conditions include but are not limited to gastroparesis and gastric bypass surgery

F. Individuals with conditions prone to hypergastrinemia (Zollinger-Ellison syndrome, use of histamine-2 receptor blockers) or hypogastrinemia (gastric surgery).

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2009-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Balow James, MD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bach JF, Chatenoud L. Tolerance to islet autoantigens in type 1 diabetes. Annu Rev Immunol. 2001;19:131-61. doi: 10.1146/annurev.immunol.19.1.131. PMID 11244033
- [Background] Lernmark A, Barmeier H, Dube S, Hagopian W, Karlsen A, Wassmuth R. Autoimmunity of diabetes. Endocrinol Metab Clin North Am. 1991 Sep;20(3):589-617. PMID 1935920
- [Background] Mathis D, Vence L, Benoist C. beta-Cell death during progression to diabetes. Nature. 2001 Dec 13;414(6865):792-8. doi: 10.1038/414792a. PMID 11742411

RESULTS

PARTICIPANT FLOW:
Groups:
- T1D Group: Subjects between the ages of 16 and 30 years, with T1D diagnosed within the preceding 6 month period, and with measurable circulating C-peptide levels.
Period: Overall Study
Arm/Group | T1D Group
Started | 7
Completed | 3
Not Completed | 4
Not completed — Protocol Violation | 3
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | T1D Group
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 6
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 21.9 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in C-peptide
Time Frame: 6 months following the protocol subject's randomization/treatment initiation
Population: Only 3 subjects completed study
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | T1D Group
Number analyzed (Participants) | 3
ng/mL | 0.51 (0.53)

2. Secondary Outcome: Glycemia Control (Change in HbA1c Level)
Time Frame: 6 months following the protocol subject's randomization/treatment initiation
Population: Only 3 subjects completed study
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | T1D Group
Number analyzed (Participants) | 3
Percentage | -1.17 (0.45)

3. Secondary Outcome: Change in Insulin Dose
Time Frame: 6 months following the protocol subject's randomization/treatment initiation
Measure: Mean (Standard Deviation); unit: U/kg/day
Arm/Group | T1D Group
Number analyzed (Participants) | 3
U/kg/day | 0.02 (0.32)

4. Secondary Outcome: Change in Anti-GAD Autoantibody Titers
Time Frame: 6 months following the protocol subject's randomization/treatment initiation
Measure: Mean (Standard Error); unit: Titers
Arm/Group | T1D Group
Number analyzed (Participants) | 3
Titers | 119278 (174649)

5. Secondary Outcome: Change in Anti-IA2 Titer
Time Frame: 6 months following the protocol subject's randomization/treatment initiation
Measure: Mean (Standard Error); unit: Titers
Arm/Group | T1D Group
Number analyzed (Participants) | 3
Titers | -29212 (49956)

6. Secondary Outcome: Change in ZnT8 Autoantibody Titer
Time Frame: 6 months following the protocol subject's randomization/treatment initiation
Measure: Mean (Standard Error); unit: Titers
Arm/Group | T1D Group
Number analyzed (Participants) | 3
Titers | -0.11 (0.19)

ADVERSE EVENTS:
Arm/Group | T1D Group
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 3/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | T1D Group (N=7)
Hypoglycemic events (Metabolism and nutrition disorders) | 3/3 (104) — According to the protocol, hypoglycemia adverse events are described as follows: Mild= BG < 65 mg/dL Moderate = BG < 54 mg/dL & symptomatic Severe = patient required assistance to obtain treatment for the event.
Rhinitis (General disorders) | 1/3 (1)
Eczema (General disorders) | 1/3 (2)
Warts (General disorders) | 1/3 (2)
Thrombocytopenia (General disorders) | 1/3 (1)
Gastroenteritis (General disorders) | 1/3 (2)
Anemia (General disorders) | 1/3 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes